CLINICAL TRIAL: NCT04505228
Title: The Personalized Chinese Herb Formulas Are Evaluated for Their Effectiveness to Relieve Symptoms in Hypertensive Bradyarrhythmia
Brief Title: The Personalized Chinese Herb Formulas Over Hypertensive Bradyarrhythmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Xiao (Other)
Collaborators: Qingdao Fifth People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Jun Xiao, Principal Investigator, Macrohard Institute of Health
Organization: Macrohard Institute of Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: qdms17337nsh
Record Dates: First submitted 2020-08-02; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Hypertensive Heart Disease
MeSH Terms: interventions — Honghua extract, Carthamus tinctorius; Immunoglobulin G; Sensitivity and Specificity; Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research group (Experimental): The patients receiving Atropine and the extra Chinese herb formulas treatment
  Interventions: Drug: Safflower (Carthamus Tinctorius) IgG4 | Serum | Allergy; Drug: Atropine Sulfate
- Control group (Active Comparator): The patients receiving the basic treatment of atropine
  Interventions: Drug: Atropine Sulfate

INTERVENTIONS:
Drug: Safflower (Carthamus Tinctorius) IgG4 | Serum | Allergy — The designed Chinese herb formulas
  Other Names: Xuefuzhuyu
  Arms: Research group
Drug: Atropine Sulfate — The basic treatment for heart disease

SUMMARY:
72 patients who have been diagnosed with hypertensive bradyarrhythmia were selected and randomly divided into research group and control group. The research group received regular medication against hypertension and the personalized formulas based on syndrome differentiation, meanwhile the control group only received the regular medication. The five symptoms (palpitation, short of breath, angina, dizzy and lumbar debility) were graded and used for evaluation of treatment.

DETAILED DESCRIPTION:
To test the effect of Chinese herb against the hypertensive heart disease, we designed this randomized controlled clinical trial. 72 patients who have been diagnosed with hypertensive bradyarrhythmia were selected and randomly divided into research group and control group. The five symptoms (palpitation, short of breath, angina, dizzy and lumbar debility) were graded. The research group received regular medication against hypertension and the personalized formulas based on syndrome differentiation, meanwhile the control group only received the regular medication. 2 weeks after treatment, all the symptoms were graded again.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertensive bradyarhhythmia

Exclusion Criteria:

* With other elementary diseases
* With pregnant
* With receiving other treatment within past half year from the beginning of trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
typical symptoms in patients with hypertensive bradyarrhythmia | 2 weeks
  The five indexes of typical symptoms in patients with hypertensive bradyarrhythmia (palpitation, angina, shortness of breath, dizzy, lumbar debility) were evaluated and scored both before treatment and after treatment according to "Guiding principles for clinical research of new Chinese Medicine".

CONTACTS AND LOCATIONS:
Locations (1):
- The fifth Qingdao people's hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided